CLINICAL TRIAL: NCT02228304
Title: A Multi-Center, Two-Stage, Open-Label Phase I and Randomized, Active Controlled, Masked Phase II Study to Evaluate the Safety and Efficacy of Intravitreal Implantation of NT-503-3 Encapsulated Cell Technology Compared With Eylea for the Treatment of Recurrent CNV Secondary to AMD
Brief Title: Study of the Intravitreal Implantation of NT-503-3 Encapsulated Cell Technology (ECT) for the Treatment of Recurrent Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After enrolling approximately 1/2 of the trial participants, the rescues exceeded stopping criteria.
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NT-503-3-AMD-001
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Macular Degeneration
Keywords: Wet AMD; Wet Age Related Macular Degeneration; Recurrent CNV Secondary to AMD; Active subfoveal CNV
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NT-503-3 ECT implantation (Experimental)
  Interventions: Drug: NT-503-3 ECT implantation
- Eylea® injected intravitreally every 8 weeks (Active Comparator): Eylea® injected intravitreally every 8 weeks
  Interventions: Drug: Eylea® injected intravitreally administered every 8 weeks

INTERVENTIONS:
Drug: NT-503-3 ECT implantation — NT-503-3 ECT implantation is a biological sustained drug delivery device that could provide continuous delivery of an anti-VEGF therapy
  Arms: NT-503-3 ECT implantation
Drug: Eylea® injected intravitreally administered every 8 weeks — The first part, stage 1, Phase I is open label with the experimental treatment arm only. Eylea® injected intravitreally is only used as a comparator in the stage 2, Phase II, portion of the study.
  Arms: Eylea® injected intravitreally every 8 weeks

SUMMARY:
Prospective, multi-center 2-stage study. Stage 1 (Phase I) is open-label with all patients treated with the NT-503-3 ECT implant. Stage 1 (Phase I) patients will undergo explantation at year 2. Those who, in the opinion of the investigator, are still candidates for continued anti-VEGF therapy will be re-implanted with a new NT-503-3 investigational product and followed for an additional 12 weeks before study exit. Stage 2 (Phase II) is a separate, randomized, masked phase during which eligible patients will be randomized to the NT-503-3 group or the control group.

Clinical Hypotheses:

* NT-503-3 ECT is comparable to Eylea® injected intravitreally every 8 weeks in the prevention of vision loss due to recurrent CNV secondary to AMD
* NT-503-3 ECT has an acceptable safety profile

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of Active (recurrent or persistent) subfoveal CNV lesions secondary to AMD in the study eye
* Prior Intravitreal Anti-VEGF injections

Key Exclusion Criteria:

* Significant subretinal hemorrhage
* Significant Scar and/or, fibrosis
* Suspected polypoidal choroidopathy, or pigment epithelial tears or rips
* Inadequate response to anti-VEGF therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with less than a 3-line loss of BCVA in ETDRS letters | Week 52 and Week 108

SECONDARY OUTCOMES:
Change from baseline in best corrected visual acuity (BCVA) | Week 52
Change from baseline in macular thickness as determined by Spectral Domain Optical Coherence Tomography (sdOCT) | Up to Week 108
Mean (median) number of Eylea® injections and number of patients requiring Eylea® injections for rescue therapy | Up to Week 108

CONTACTS AND LOCATIONS:
Overall Officials: Charles Johnson, MB, ChB, Study Chair — Neurotech Pharmaceuticals, Inc.
Locations (38):
- United States (32):
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California, Irvine, The Gavin Herbert Eye Institute, Irvine, California
  - Jacobs Retina Center at UCSD, La Jolla, California
  - Colorado Retina Associates, Golden, Colorado
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Georgina Retina, P.C., Marietta, Georgia
  - Illinois Retina Associates, S.C., Joliet, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Retina Associates of Kentucky, Lexington, Kentucky
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, PC, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - William Beaumont Hospital-Ophthalmology Research, Royal Oak, Michigan
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, LLC, Bloomfield, New Jersey
  - NJ Retina, New Brunswick, New Jersey
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Palmetto Retina Center, LLC, Florence, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Hadassah-Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center,, Tel Aviv